CLINICAL TRIAL: NCT03429972
Title: Regional Cryotherapy in Preventing Paclitaxel Induced Peripheral Neuropathy in Patients With Early and Locally Advanced Breast Cancer
Brief Title: Regional Cryotherapy in Preventing Paclitaxel Induced Peripheral Neuropathy in Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Terry Fox Foundation (Other); Duke-NUS Academic Medicine Research Institute (Unknown); Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015/3017
Record Dates: First submitted 2017-11-09; First posted 2018-02-12 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: Paclitaxel; Neuropathy
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paclitaxel and Elasto-Gel™ Cryotherapy (Experimental): Cryotherapy will be applied using Elasto-Gel™ hypothermia mitts and slippers for 15 minutes before, during and 15 minutes after each paclitaxel infusion.
  Interventions: Device: Elasto-Gel™; Drug: Paclitaxel
- Paclitaxel alone (Other): Paclitaxel will be administered without cryotherapy.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Device: Elasto-Gel™ — Elasto-Gel™ hypothermia mitts and slippers contain glycerine, which has thermal properties, allowing use for cold therapies.
  Arms: Paclitaxel and Elasto-Gel™ Cryotherapy
Drug: Paclitaxel — 80mg/m^2 of Paclitaxel is administered by infusion for 60 mins once a week, for a total of 12 cycles

SUMMARY:
The trial will be preceded by a pilot phase study in 5 patients.

This will then be followed by the randomized 1:1 phase II trial testing the utility of regional cryotherapy in preventing or reducing paclitaxel-induced peripheral neuropathy compared to no treatment.

It is hypothesized that cryotherapy causes regional blood vessel constriction and decreases the paclitaxel exposure to the distal epithelial nerve fibres, thus resulting in decreased nerve damage.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent prior to any study specific procedures.
2. Age ≥ 21 years old
3. Patients with histologically confirmed early or locally advanced breast cancer
4. Must be receiving 12x weekly sessions of paclitaxel as part of their adjuvant or neo-adjuvant chemotherapy
5. Must have routine chemotherapy lab investigations as per institutional practice
6. Concurrent use of Trastuzumab and/or Pertuzumab for cerbB-2 positive patients as per institutional practice is allowed
7. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.

Exclusion Criteria:

1. Patients diagnosed with pre-existing or history of peripheral neuropathy (regardless of cause)
2. Patients with history of Raynaud's disease
3. Prior use of taxane-based chemotherapy
4. Concurrent use of other neuro-toxic chemotherapy with paclitaxel
5. Patients who have had any axillary clearance surgery and without a central venous access device for chemotherapy administration
6. Patients with any severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate patient participation in the clinical study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients reporting level C and above subjective symptoms, in cryotherapy arm versus controlled arm, based on the Patient Neurotoxicity Questionnaire (PNQ) at 3 months after baseline | From commencement to completion of 12 paclitaxel infusions - estimated 3 months
  PNQ scale ranges from scores A to E; with scoring of A being not affected neuropathy, and E with the worst neuropathy

SECONDARY OUTCOMES:
Proportion of patients reporting level C and above subjective symptoms, in cryotherapy arm versus controlled arm, based on the Patient Neurotoxicity Questionnaire (PNQ) at 15 months after baseline | From commencement to completion of primary chemotherapy - estimated 15 months
Proportion of patients with lower sensory velocity and amplitudes (based on nerve conduction tests), in cryotherapy arm versus controlled arm, at 15 months after baseline | From commencement to completion of primary chemotherapy - estimated 15 months
Incidence of adverse events, in cryotherapy arm versus controlled arm | From commencement to completion of 12 paclitaxel infusions - estimated 3 months
Proportion of patients reported intolerance and require cessation of therapies, in cryotherapy arm versus controlled arm | From commencement to completion of 12 paclitaxel infusions - estimated 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kiley Loh Wei-Jen, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ng DQ, Tan CJ, Soh BC, Tan MML, Loh SY, Tan YE, Ong HH, Teng PPC, Chan JJ, Chay WY, Lee J, Lai G, Beh SY, Tan TJY, Yap YS, Lee GE, Wong M, Dent R, Lo YL, Chan A, Loh KW. Impact of Cryotherapy on Sensory, Motor, and Autonomic Neuropathy in Breast Cancer Patients Receiving Paclitaxel: A Randomized, Controlled Trial. Front Neurol. 2020 Dec 18;11:604688. doi: 10.3389/fneur.2020.604688. eCollection 2020. PMID 33424755